CLINICAL TRIAL: NCT04714684
Title: The Role of Fitostimoline Proctogel in Symptoms Relief and Healing in Patients Affected by Anal Fissure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Gian Luca Baiocchi, Prof., Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FITOSTIMOLINE
Record Dates: First submitted 2020-11-27; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Fissure in Ano
MeSH Terms: conditions — Fissure in Ano

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- fitostimoline proctogel (Experimental)
  Interventions: Device: Fitostimoline proctogel; Device: Fitostimoline proctogel + muscle relaxant
- fitostimoline proctogel + muscle relaxants (Experimental)
  Interventions: Device: Fitostimoline proctogel; Device: Fitostimoline proctogel + muscle relaxant
- muscle relaxants (Experimental)
  Interventions: Device: Fitostimoline proctogel; Device: Fitostimoline proctogel + muscle relaxant

INTERVENTIONS:
Device: Fitostimoline proctogel — Medical device for topical use for the treatment of fissures
  Other Names: muscle relaxant
Device: Fitostimoline proctogel + muscle relaxant — medical device for topical use for the treatment of fissures

SUMMARY:
Evaluate the effectiveness of fitostimoline proctogel in the anal fissure healing and in the need for invasive interventions (primary endpoints) and in the healing of the fissure (secondary endpoint) using Fitostimoline in addition to or without other topical devices available on the market.

Three groups will be established: one for the exclusive use of fitostimoline, the second for the use of fitostimoline in addition to one of the other topical devices already on the market and the third group only for the use of other topical therapies.

ELIGIBILITY:
Inclusion Criteria:

* None previous therapies for anal fissure
* Symptomatic anal fistula
* Signing of informed consent
* age >18 years old

Exclusion Criteria:

* Patients unable to complete the questionnaire and with a legal guardian.
* Patients with concomitant abscess/fistula
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-10 (Estimated); Primary Completion 2022-02-10 (Estimated); Study Completion 2022-02-10 (Estimated)

PRIMARY OUTCOMES:
control of anal fissure symptoms | 30 days
  pain relief (by using the NRS scale from 0 to 10 (0=absence of pain 10= maximum presence of pain) which should be lower than 3)
need of invasive treatment | 30 days
  Anal dilatation, lateral internal sphincterotomy

SECONDARY OUTCOMES:
anal fissure healing | 30 days
  no pain (NRS scale < 1, where 0 is absence of pain and 10 is maximum pain), no bleeding